CLINICAL TRIAL: NCT00589420
Title: A Phase II Study of Sorafenib in Combination With Docetaxel in Patients With Androgen-Independent Prostate Cancer
Brief Title: Sorafenib and Docetaxel in Patients With Prostate Cancer That Did Not Respond to Previous Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Sanofi (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03806; 805372 (Other: University of Pennsylvania IRB); CDR0000581020 (Other: Sanofi)
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Phase II (Experimental): All patients received sorafenib 200 mg bid daily and docetaxel 75 mg/m2 every 3 weeks
  Interventions: Drug: docetaxel; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: docetaxel
  Other Names: Taxotere
Drug: sorafenib tosylate
  Other Names: Nexavar

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with docetaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying giving sorafenib together with docetaxel to see how well it works in treating patients with metastatic androgen-independent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of patients achieving a 50% reduction in serum PSA from baseline in patients with androgen-independent prostate cancer (AIPC) receiving sorafenib tosylate and docetaxel.

Secondary

* To estimate the progression-free survival of patients with AIPC.
* To quantify the number and percent of patients who have stable disease at 6 months of therapy (failure to progress).
* To estimate median time to progression for all patients.
* To estimate the objective response rate of patients with AIPC treated with this regimen.
* To measure the percentage of patients surviving at 2 years.
* To determine the toxicities and estimate toxicity rates for patients treated with this regimen.
* To measure changes in tumor vasculature in response to therapy in selected patients with dynamic contrast-enhanced MRI (DCE-MRI) and correlate primary and secondary objectives to these measurement changes.
* To measure changes in serum HMGB1 in response to therapy and correlate primary and secondary objectives with these changes.
* To measure changes in serum cathepsin D in response to therapy and correlate primary and secondary objectives with these changes.

OUTLINE: Patients receive oral sorafenib tosylate twice daily on days 2-19 and docetaxel IV on day 1. Treatment repeats every 21 days for up to 10 courses. Patients then receive oral sorafenib tosylate alone twice daily on days 1-19 with treatment repeating every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically to measure serum HMGB1 and cathepsin D levels before and after therapy.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate with clinical or radiological evidence of metastatic disease.
* Serum PSA >5 ng/mL.
* Patients must have discontinued flutamide or nilutamide for at least 4 weeks and bicalutamide for at least 6 weeks
* Disease progression during hormonal therapy defined as at least one of the following:

  1. increasing serum PSA levels on at least two measurements at least two weeks apart.
  2. Progressive measurable disease (by RECIST criteria) independent of PSA
  3. Bone scan progression with at least one new lesion.
* Serum testosterone ≤ 50 ng/dL. Patients must be receiving primary androgen ablation therapy with a GnRH agonist as maintenance therapy unless surgically castrated.
* Age > 18 years.
* ECOG performance status of ≤ 1.
* Baseline laboratory values (evaluated within 14 days of randomization):

White Blood Count > 3,000/mm3 Absolute Granulocyte Count > 1,500/mm3 Platelet Count > 100,000/mm3 Serum creatinine < 2.0 x upper limit of normal (ULN) INR < 1.5 before the start of chronic anticoagulation and a PTT within normal limits

* Liver Function Total Bilirubin less or equal to ULN AST and ALT must be <5X ULN for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used.
* Prior radiation therapy is allowed. However, if radiation has been administered to a lesion, there must be radiographic evidence of progression of that lesion in order for that lesion to constitute measurable disease or to be included in the measured target lesions. 4 weeks must have elapsed between radiation therapy and entry into study.
* Prior vaccine therapy is allowed
* Prior and/or concurrent zoledronic acid (Zometa) therapy is allowed.
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion criteria:

* Prior therapy with cytotoxic chemotherapy
* Prior therapy with radioisotopes
* History of brain metastasis or leptomeningeal disease
* Symptomatic neuropathy >grade2
* Prior history of cancer (except basal cell or squamous-cell skin cancer) within the past 5 years (exceptions must be approved by the PI)
* Prior history of DVT or Pulmonary embolism in the last 1 year
* Patients must not have a serious medical illness including, but not limited to, ongoing or active infection requiring parental antibiotics; clinically significant cardiovascular disease (e.g. uncontrolled hypertension, recent myocardial infarction, unstable angina), New York heart association grade II or greater congestive heart failure, or grade II or greater peripheral arterial vascular within 1 year prior to study entry, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), rifampin or St. John's wort.
* Patients must not be taking drugs that inhibit CYP3A at the time of enrollment to prevent drug-drug interactions with docetaxel. These include ketoconazole, voriconazole, itraconazole, fluconazole, cimetidine, clarithromycin, erythromycin, troleandomycin, and grapefruit juice. These agents should be avoided during treatment while on study.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with bone marrow-suppressive therapy, HIV-positive patients are excluded from the study. For patients receiving combination anti-retroviral therapy, the potential impact of pharmacokinetic interactions with sorafenib and docetaxel is unknown. Appropriate studies may be undertaken in patients with HIV and those receiving combination anti-retroviral therapy in the future.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07-27 (Actual); Primary Completion 2010-02-02 (Actual); Study Completion 2011-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, RN, MPA, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD will be done on a case by case basis

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II Trial of Sorafenib and Docetaxel: All patients received sorafenib 200 mg bid daily and docetaxel 75 mg/m2 every 3 weeks
  docetaxel
  sorafenib tosylate
Period: Overall Study
Arm/Group | Phase II Trial of Sorafenib and Docetaxel
Started | 18
Completed | 17
Not Completed | 1
Not completed — screen failure | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients that received both drugs
Groups:
- Sorafenib and Docetaxel: All patients received sorafenib 200 mg bid daily and docetaxel 75 mg/m2 every 3 weeks
  docetaxel
  sorafenib tosylate
Arm/Group | Sorafenib and Docetaxel
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: PSA Response: ≥50% decline from baseline PSA measurement confirmed by a second PSA measurement 3 weeks later. Patients may not demonstrate clinical or radiographic evidence of disease progression.
  PSA progression (PSA-P): Two measurements of rising serum PSA measured at least 2 weeks apart where the second is greater than the first.
Time Frame: From start of treatment until withdrawal from the study, approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Trial of Sorafenib and Docetaxel
Number analyzed (Participants) | 17
Participants | 6

2. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: Number of patients that achieved 6 month PFS
Time Frame: 6 months from end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Trial of Sorafenib and Docetaxel
Number analyzed (Participants) | 17
Participants | 10

3. Secondary Outcome: Objective Response Rate (ORR)
Description: To determine the ORR in patients with measurable disease
Time Frame: 6 months from end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Trial of Sorafenib and Docetaxel
Number analyzed (Participants) | 18
Participants | 3

ADVERSE EVENTS:
Time Frame: first treatment through study completion, approximately 12 months
Arm/Group | Phase II Trial of Sorafenib and Docetaxel
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Trial of Sorafenib and Docetaxel (N=17)
anemia (Blood and lymphatic system disorders) | 3 (3)
anorexia (Metabolism and nutrition disorders) | 1 (1)
diarreha (Gastrointestinal disorders) | 1 (1)
fatigue (Metabolism and nutrition disorders) | 3 (3)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
hypertension (Cardiac disorders) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 5 (5)
nausea (Gastrointestinal disorders) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 17 (17)
pneumonia (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Weight Loss (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes